CLINICAL TRIAL: NCT05894096
Title: Air Cold Atmospheric Pressure Plasma Treatment for Acceleration of Venous Ulcer Healing
Acronym: PLASFRI-CUV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Complejo Hospitalario La Mancha Centro (Other); FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLASFRI-CUV
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Venous Leg Ulcer
Keywords: Cold atmospheric plasma; venous ulcer; wound healing
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: * Prospective, randomized, open-label, controlled clinical trial with conventional treatment.
  * Programming and continuous recruitment.
  * The ulcers of the experimental group will be treated with 60 seconds/cm2 of the wound surface, carried out twice a week, and with alginate with silver. For their part, the ulcers in the control group will be treated with alginate with silver, which will also be replaced twice a week.
  * The total duration of the trial for each patient will be 10 weeks (2 times per week) followed by 8 weeks of follow-up.
  * The treatment will be carried out twice a week, maintaining at least 72 hours between treatments.
  * The patients included in this trial will be all those who attend consultations or are hospitalized. They must present at least one venous ulcer larger than 1 cm2 that has not healed in the last 8 weeks from its onset and with no surgical indication for ulcer coverage by a skin graft.
Who Masked: Participant
Masking Description: Patients will be randomly distributed into two arms: Experimental and Control. Ulcers will be treated in all patients of the experimental arm using the PlasmAction Med cold plasma generator. The plasma jet will be programmed to be applied with an intensity of 55% power and with 60 seconds/cm2 of surface, the frequency being twice a week for 10 weeks. This therapeutic regimen is based on previous studies of previously published clinical trials with argon jet cold plasma (14,15). The administration of treatment will be the responsibility of the principal investigator and the collaborator with the help of the nursing staff. After the application of the plasma treatment, the patient will then be cured with alginate (Melgisorb Ag®) of the size 10 X 10 cm and 5x5 (3 units). For patients included in the control arm, alginate (Melgisorb Ag®) will be used as a cure for ulcers, size 10 X 10 cm and 5x5 (3 units), whose replacements will also be carried out twice a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold Athmospheric Plasma Jet+Alginate patch (Experimental): Leg Venous Ulcers will be treated in all patients belonging to the experimental arm using the PlasmAction Med cold plasma generator at atmospheric air pressure and alginate (Melgisorb Ag®) will be used after the plasma has been applied.
  Interventions: Device: Cold Atmospheric Plasma Jet Treatment; Device: Alginate Patch
- Alginate patch (Active Comparator): For patients included in the control arm, alginate (Melgisorb Ag®) will be used as a cure for ulcers, size 10 X 10 cm and 5x5 (3 units), whose replacements will also be carried out twice a week.
  Interventions: Device: Alginate Patch

INTERVENTIONS:
Device: Cold Atmospheric Plasma Jet Treatment — Application of Colf Atmospheric Plasma Jet on the wound
  Arms: Cold Athmospheric Plasma Jet+Alginate patch
Device: Alginate Patch — Application of Alginate Patches on the wound

SUMMARY:
In this medical trial, a novel prototype of a medical device based on a Cold Atmospheric Air Plasma Jet for the treatment is clinically tested on patients with venous leg ulcers. The device is characterized by producing the first cold air plasma jet compatible with living tissues at a low heat transfer rate with a temperature on the skin surface lower than 40 ºC. It has a practical design to be used by physicians during daily practice with a special focus on unhealed ulcers.

DETAILED DESCRIPTION:
The device to be validated in this test is an air-generating unit in a cold plasma state, a prototype of a medical device. Cold plasma-generating equipment is already available on the market and is intended for the treatment of chronic ulcers in patients. Its technology is based on the generation of a plasma jet produced with the noble gas argon. The novelty of this new plasma generator lies in the fact that its production is carried out by using atmospheric air, which implies greater efficiency and ease of use, being the first of its kind at an international level. The main mechanism of action underlying the therapeutic effect of cold atmospheric plasmas is the effect of the electric fields produced by the charged particles that make up the air in the plasma state. These fields are imperceptible to the patient, however, the effect on microcirculation in the area of application of the wound is very noticeable. The improvement in microcirculation extends for a longer time than the treatment as demonstrated by reported oxygen saturation studies using cold air plasmas DBD (Dielectric Barrier Discharge) that include clinical trials (1-4). Enhanced capillary blood flow increases local oxygen saturation and nutrient supply, thus promoting wound healing (5). In addition to the action of electric fields, there is an auxiliary decontamination mechanism generated by the emission of ultraviolet radiation, below the damage threshold for humans and excited and ionized oxygen and nitrogen molecules. This mechanism eliminates bacteria, including resistant ones, so that the regeneration capacity promoted by the main mechanism of action is enhanced (6-8).

The generator chosen for this test belongs to the Spanish company ION BIOTEC S.L. (PlasmAction Med), which has obtained an international patent (9). Its use in animals has been successfully developed in veterinary clinics and the positive results obtained in the closure of torpid ulcers using cold atmospheric plasmas have been demonstrated (10-13). The plasma jet is applied directly to the lesion presented by the patient with a power of 55% and with an intensity and duration of 60 s/cm2, by means of the regulator found at the end of an application hose. It does not use consumables or produce waste.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (18 years).
* Signed informed consent.
* Presenting at least one venous ulcer larger than 1 cm2 that has not healed in the last 3 weeks from its appearance.
* Absence of surgical indication for ulcer coverage by skin graft.

Exclusion Criteria:

* Uncontrolled diabetes mellitus (HbA1c > 8%). If during the trial the patient suffers a decompensation of diabetes, it will be considered an adverse event.
* Patient allergic to silver or any other material that will be used during the cure of the ulcer under study.
* Concomitant treatment with vacuum-assisted closure (VAC) therapy.
* Use of topical antibiotic therapy. The minimum washing time should be 48 hours.
* Presence of critical limb ischemia defined as an ankle-brachial index (ABI) below 0.5 or a transcutaneous O2 pressure (TcPO2) below 15 mmHg.
* Treatment with corticosteroids in the 14 days prior to the study or with other immunosuppressants.
* Presence of a chronic or active skin disorder that may negatively influence wound healing (such as Marfan or Ehlers-Danlos syndrome, systemic lupus erythematosus, systemic sclerosis, or psoriasis).
* Pregnancy or lactation.
* Advanced or metastatic stage cancer.
* Deficiency states.
* Dementia.
* Post radiation wounds.
* Sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer Surface | 18 weeks
  The surface of the ulcer will be meassured by means of sofware image J2

SECONDARY OUTCOMES:
Measurement of bacterial burden | 18 weeks
  Bacteriological cultures will be taken before and after of the treated group at 0, 5 and 10 weeks. Control groups at º, 5 and 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo C Hontanilla, Ph.D., Study Director — Clínica Universidad de Navarra; José M Lasso Vázquez, Ph.D., Principal Investigator — Hospital General Universitario Gregorio Marañón; Jesús J Castellanos Monedero, M.D., Principal Investigator — Hospital General la Mancha-Centro; Javier Buendía Pérez, Ph.D., Principal Investigator — Hospital San Carlos, Madrid; José I Leal Lorenzo, Ph.D., Principal Investigator — Clínica Universidad de Navarra
Locations (5):
- Spain (5):
  - Hospital General La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Clinica Universidad de Navarra, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
When finished the protocol the data collected will be shared with other researches in order to continue other clinical trials
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available in 2025 and will be availabe for 10 years

REFERENCES:
- [Background] Kisch T, Schleusser S, Helmke A, Mauss KL, Wenzel ET, Hasemann B, Mailaender P, Kraemer R. The repetitive use of non-thermal dielectric barrier discharge plasma boosts cutaneous microcirculatory effects. Microvasc Res. 2016 Jul;106:8-13. doi: 10.1016/j.mvr.2016.02.008. Epub 2016 Mar 2. PMID 26944583
- [Background] Kisch T, Helmke A, Schleusser S, Song J, Liodaki E, Stang FH, Mailaender P, Kraemer R. Improvement of cutaneous microcirculation by cold atmospheric plasma (CAP): Results of a controlled, prospective cohort study. Microvasc Res. 2016 Mar;104:55-62. doi: 10.1016/j.mvr.2015.12.002. Epub 2015 Dec 3. PMID 26655582
- [Background] Jensen JO, Schulz L, Schleusser S, Matzkeit N, Stang FH, Mailaender P, Kraemer R, Kleemann M, Deichmann H, Kisch T. The repetitive application of cold atmospheric plasma (CAP) improves microcirculation parameters in chronic wounds. Microvasc Res. 2021 Nov;138:104220. doi: 10.1016/j.mvr.2021.104220. Epub 2021 Jun 30. PMID 34216601
- [Background] Matzkeit N, Schulz L, Schleusser S, Jensen JO, Stang FH, Mailaender P, Kramer R, Kisch T. Cold atmospheric plasma improves cutaneous microcirculation in standardized acute wounds: Results of a controlled, prospective cohort study. Microvasc Res. 2021 Nov;138:104211. doi: 10.1016/j.mvr.2021.104211. Epub 2021 Jun 16. PMID 34144075
- [Background] Heuer K, Hoffmanns MA, Demir E, Baldus S, Volkmar CM, Rohle M, Fuchs PC, Awakowicz P, Suschek CV, Oplander C. The topical use of non-thermal dielectric barrier discharge (DBD): nitric oxide related effects on human skin. Nitric Oxide. 2015 Jan 30;44:52-60. doi: 10.1016/j.niox.2014.11.015. Epub 2014 Nov 27. PMID 25435001
- [Background] MORFILL G. TREATING DEVICE FOR TREATING A BODY PART OF A PATIENT WITH A NON-THERMAL PLASMA. WO 2010/094307 Al, 2009.
- [Background] Ziuzina D, Boehm D, Patil S, Cullen PJ, Bourke P. Cold Plasma Inactivation of Bacterial Biofilms and Reduction of Quorum Sensing Regulated Virulence Factors. PLoS One. 2015 Sep 21;10(9):e0138209. doi: 10.1371/journal.pone.0138209. eCollection 2015. PMID 26390435
- [Background] Cooper M, Fridman G, Fridman A, Joshi SG. Biological responses of Bacillus stratosphericus to floating electrode-dielectric barrier discharge plasma treatment. J Appl Microbiol. 2010 Dec;109(6):2039-48. doi: 10.1111/j.1365-2672.2010.04834.x. PMID 20825520
- [Background] CORTÁZAR PÉREZ OD, MEGIA MACÍAS AM. Electromedical device for blood clotting and treatment of ulcers and other skin injuries in human and animal patients. 2020.
- [Background] Ulrich C, Kluschke F, Patzelt A, Vandersee S, Czaika VA, Richter H, Bob A, Hutten Jv, Painsi C, Huge R, Kramer A, Assadian O, Lademann J, Lange-Asschenfeldt B. Clinical use of cold atmospheric pressure argon plasma in chronic leg ulcers: A pilot study. J Wound Care. 2015 May;24(5):196, 198-200, 202-3. doi: 10.12968/jowc.2015.24.5.196. PMID 25970756
- [Background] Chuangsuwanich A, Assadamongkol T, Boonyawan D. The Healing Effect of Low-Temperature Atmospheric-Pressure Plasma in Pressure Ulcer: A Randomized Controlled Trial. Int J Low Extrem Wounds. 2016 Dec;15(4):313-319. doi: 10.1177/1534734616665046. Epub 2016 Sep 20. PMID 27581113
- [Background] A. Nishijima. A New Energy Device for Skin Activation to Acute Wound Using Cold Atmospheric Pressure Plasma: A Randomized Controlled Clinical Trial. Biomed J Sci Tech Res. 2019;21(1):15494-501. DOI: 10.26717/BJSTR.2019.21.003532
- [Background] Amini MR, Sheikh Hosseini M, Fatollah S, Mirpour S, Ghoranneviss M, Larijani B, Mohajeri-Tehrani MR, Khorramizadeh MR. Beneficial effects of cold atmospheric plasma on inflammatory phase of diabetic foot ulcers; a randomized clinical trial. J Diabetes Metab Disord. 2020 Jul 14;19(2):895-905. doi: 10.1007/s40200-020-00577-2. eCollection 2020 Dec. PMID 33520811
- [Background] Brehmer F, Haenssle HA, Daeschlein G, Ahmed R, Pfeiffer S, Gorlitz A, Simon D, Schon MP, Wandke D, Emmert S. Alleviation of chronic venous leg ulcers with a hand-held dielectric barrier discharge plasma generator (PlasmaDerm((R)) VU-2010): results of a monocentric, two-armed, open, prospective, randomized and controlled trial (NCT01415622). J Eur Acad Dermatol Venereol. 2015 Jan;29(1):148-55. doi: 10.1111/jdv.12490. Epub 2014 Mar 25. PMID 24666170
- [Background] Brany D, Dvorska D, Halasova E, Skovierova H. Cold Atmospheric Plasma: A Powerful Tool for Modern Medicine. Int J Mol Sci. 2020 Apr 22;21(8):2932. doi: 10.3390/ijms21082932. PMID 32331263